CLINICAL TRIAL: NCT03900104
Title: Cervical and Endometrial Injection for Sentinel Lymph Node Detection in Endometrial Cancer: A Prospective Randomized Trial
Brief Title: Cervical and Endometrial Injection for Sentinel Lymph Node Detection in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CEIN
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node
Keywords: Endometrial Cancer; Sentinel Lymph Node; Paraaortic nodes involvement
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcervical endometrial injection arm (Experimental): Tracer injection performed by a transcervical catheter in endometrial cancer patients.
  Interventions: Procedure: Transcervical endometrial injection of technetium 99 m-labeled human albumin colloid particles
- Cervical injection arm (Active Comparator): Tracer injection was administered via the cervical route in endometrial cancer patients.
  Interventions: Procedure: Cervical injection of technetium 99 m-labeled human albumin colloid particles

INTERVENTIONS:
Procedure: Transcervical endometrial injection of technetium 99 m-labeled human albumin colloid particles — Transcervical endometrial injection of technetium 99 m-labeled human albumin colloid particles, in 5 mL saline, 2 hours before surgery. Injection performed with a trans-cervical catheter
  Arms: Transcervical endometrial injection arm
Procedure: Cervical injection of technetium 99 m-labeled human albumin colloid particles — Cervical injection of technetium 99 m-labeled human albumin colloid particles, in 5 mL saline, 2 hours before surgery.
  Arms: Cervical injection arm

SUMMARY:
The investigators think that trans-cervical endometrial tracer injection will cause more paraaortic sentinel lymph node detection. Also, this application is easy, cost-effective and safer than hysteroscopic method. Transtubal tumor spearing will not occur with this method.

DETAILED DESCRIPTION:
Endometrial tracer injection will be performed by cervical or transcervical endometrial methods. Pelvic and para-aortic sentinel lymph node detection capacity will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial Cancer Patients
* Suitable patients for surgical staging

Exclusion Criteria:

* Patients who cannot undergo cervical or transcervical endometrial injection
* Pathology did not confirm endometrial cancer
* Sarcoma of the uterine corpus
* If a 90-day follow-up was not feasible

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Detected pelvic and paraaortic sentinel lymph node numbers | Postoperative 30 days
  Detected pelvic and paraaortic sentinel lymph node numbers in pathological examination (Ultrastaging)

SECONDARY OUTCOMES:
Numbers adverse events | Postoperative 90 days
  Number of adverse events associated with the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Şener Gezer, M.D, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solima E, Martinelli F, Ditto A, Maccauro M, Carcangiu M, Mariani L, Kusamura S, Fontanelli R, Grijuela B, Raspagliesi F. Diagnostic accuracy of sentinel node in endometrial cancer by using hysteroscopic injection of radiolabeled tracer. Gynecol Oncol. 2012 Sep;126(3):419-23. doi: 10.1016/j.ygyno.2012.05.025. Epub 2012 May 30. PMID 22659192
- [Background] Niikura H, Kaiho-Sakuma M, Tokunaga H, Toyoshima M, Utsunomiya H, Nagase S, Takano T, Watanabe M, Ito K, Yaegashi N. Tracer injection sites and combinations for sentinel lymph node detection in patients with endometrial cancer. Gynecol Oncol. 2013 Nov;131(2):299-303. doi: 10.1016/j.ygyno.2013.08.018. Epub 2013 Aug 27. PMID 23988415